CLINICAL TRIAL: NCT02993679
Title: Biomechanical Assessment of the Reconstruction of the Anterolateral Ligament During ACL Surgery. The In-vivo Study
Brief Title: Stability of the Knee Joint After Anterior Cruciate Ligament and Anterolateral Ligament Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Znojmo (Other)
Responsible Party: Principal Investigator, Komzak Martin, M.D., General Hospital Znojmo, Hospital Znojmo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Hospital Znojmo
Record Dates: First submitted 2016-12-04; First posted 2016-12-15 (Estimated); Last update posted 2016-12-15 (Estimated); Status verified 2016-12

CONDITIONS: Cruciate Ligament Rupture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- double-bundle ACL reconstruction (Other): surgical reconstruction of the anterior cruciate ligament
  Interventions: Procedure: reconstruction of the ACL and anterolateral ligament
- anterolateral ligament reconstruction (Other): surgical reconstruction of the anterolateral ligament
  Interventions: Procedure: reconstruction of the ACL and anterolateral ligament

INTERVENTIONS:
Procedure: reconstruction of the ACL and anterolateral ligament — reconstruction of the ACL and anterolateral ligament

SUMMARY:
The objective of this randomised cohort study was to evaluate the knee rotational stability after the single-bundle ACL reconstruction (SB) with addition of the ALL reconstruction and to compare it with the double-bundle ACL reconstruction technique (DB) and to analyse when the ALL is necessary to reconstruct.

DETAILED DESCRIPTION:
Background Rotational instability after the anterior cruciate ligament (ACL) injury and subsequent reconstruction may be caused by the rupture of the anterolateral structures of the knee, specifically the anterolateral ligament (ALL).

There are more techniques to improve the rotational stability of the knee. The objective of this randomised cohort study was: (1) To evaluate the knee rotational stability after the single-bundle ACL reconstruction (SB) with addition of the ALL reconstruction and to compare it with the double-bundle ACL reconstruction technique (DB). (2) To analyse when the ALL is necessary to reconstruct.

Methods 60 patients underwent the ACL reconstruction with the average age of 29.5 years. In thirty patient's knees the ACL was replaced with quadriceps muscle graft using the SB technique in combination with the ALL reconstruction by the gracilis graft (ALL group). With another thirty patients the ACL was reconstructed performing DB technique with the use of hamstring tendons (DB group). The rotational stability was studied before and after the reconstruction of the ACL in time "zero" using the computer navigation system. In the ALL group, the rotational stability was also analysed after the ALL reconstruction.

ELIGIBILITY:
Inclusion Criteria:

* The isolated ACL lesion
* The absence of the previous surgery on the knee joint
* The body mass index (BMI) less than 30.

Exclusion Criteria:

* Associated injuries of the tissue around the knee joint

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2014-07; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Description of the change in the rotational stability of the knee joint after ACL and anterolateral ligament reconstruction. | 24 months after the operation
  Analyse of the rotational stability of the knee joint 24 months after the operation by the computerised navigation system.

IPD SHARING:
Plan to Share IPD: Undecided